CLINICAL TRIAL: NCT01744470
Title: Efficacy and Safety Outcome of Two Different Targets of Advagraf® Trough Levels Between 4 Months and 12 Months After Transplantation Among de Novo Renal Transplant Recipients.
Brief Title: Efficacy and Safety Study of a 4-Month Post-Renal Transplant Dose Reduction of Tacrolimus(ADEQUATE)
Acronym: ADEQUATE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Tours (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHAO2011/YL/ADEQUATE; 2011-003184-29 (EudraCT Number)
Record Dates: First submitted 2012-06-11; First posted 2012-12-06 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: De Novo Transplant Disease
Keywords: Renal; Transplantation; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A - tacrolimus half-dose (Experimental): Immunosuppressive strategy with 50 % reduction of Advagraf® daily dose at M4 (randomization) and unchanged MMF dose. Targeted tacrolimus trough level are to be higher than 3 ng/mL . If the dose is not in adequation with the dispensable units, the prescribed dose will be the closest higher dose.
  Drug: Tacrolimus targeted half-dose
  Interventions: Drug: Tacrolimus targeted half-dose
- Group B - tacrolimus unchanged dose (Experimental): Immunosuppressive strategy will remain identical after randomization (M4): unchanged Advagraf® and MMF doses. Targeted tacrolimus trough level are to be between 7 and 12 ng/mL Drug: Tacrolimus targeted plain dose
  Interventions: Drug: Tacrolimus targeted plain dose

INTERVENTIONS:
Drug: Tacrolimus targeted half-dose
  Other Names: Advagraf®
  Arms: Group A - tacrolimus half-dose
Drug: Tacrolimus targeted plain dose
  Other Names: Advagraf®
  Arms: Group B - tacrolimus unchanged dose

SUMMARY:
This prospective, interventional, open label, randomized, multicenter study was designed to determine the risk/benefit ratio of a 50 % reduction of Advagraf® daily dose, 4 months after transplantation. Randomized patients are to be stable with their tacrolimus daily dose required to reach targeted tacrolimus trough levels. Based on Month-3 eligibility assessments, patients will be randomized in two groups (1:1): patients with 50 % reduction of the daily dose of Advagraf® 4 months after transplantation, and patients kept on their usual dose. The benefit/risk ratio will include the assessment of renal function, histological lesions from both alloreactivity and CNI nephrotoxicity, and safety data (metabolic and infectious diseases).

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 et 70 years
* Patient accepting to give a written informed consent
* Recipients of a first renal allograft
* Cadaver or living transplantation or living (non HLA identical) donor with compatible ABO blood type.
* Absence of positive DSA using Luminex®, MFI>1,000
* Negative cross-match in cytotoxicity
* Patient without difficulty to understand and communicate with the investigator and his collaborators
* Patient entitled to Health System benefits or other such benefits.

Exclusion Criteria:

* Multiple organ transplantation
* Recipients of a dual kidney transplant
* Previous renal allograft
* History of any other transplantation
* Receiving a graft from a non-heart-beating donor
* Patient BMI > 35
* Patients with evidence of severe liver disease, including abnormal liver profile (AST, ALT, or total bilirubin > 3 times upper limit of normal) at screening.
* Significant severe infection, active peptic ulcer and/or difficulty to absorb oral drugs (active upper gastro-intestinal tract malabsorption syndrome)
* HIV-positive patients, or with an active B or C hepatitis
* Patients with de novo malignancy prior to transplantation, other than efficiently treated basal or squamous cell carcinoma of the skin.
* Leucocyte count lower than 2500/mm3
* Female patients who are pregnant, lactating or of child bearing potential and not practicing an approved method of birth control.
* Known allergy or intolerance to basiliximab, tacrolimus, macrolide antibiotics, corticosteroids, or mycophenolate mofetil or any of the product excipients
* Participation in a clinical trial or expanded access trial with an investigational drug within 4 weeks prior to enrollment or concomitantly with this study
* Any clinical condition which, in the opinion of the investigator, would not allow safe completion of the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2012-05; Primary Completion 2015-03 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Renal function at one year post transplantation | 12 months
  Renal function at one year post transplantation estimated by the glomerular filtration rate (GFR) using MDRD 4 (Modification Diet in Renal Disease). Crude difference in renal function at one year between groups and the change of renal function between 4 months and one year in each group will be analyzed and compared.

SECONDARY OUTCOMES:
To determine and compare according to randomized group | 12 months
  Routine graft histology at M12 assessed using Banff 2009 classification, with specific analysis of interstitial fibrosis (IF) using numeric quantification
To determine and compare according to randomized group | 12 months
  Glucose metabolism at M4 and M12
To determine and compare according to randomized group | 12 months
  Infection rate including BKV and CMV at M4 and M12
To determine and compare according to randomized group | 12 months
  Presence and intensity of Donor Specific Antibody (DSA) at M3 and M12
To determine and compare according to randomized group | 12 months
  Incidence of biopsy proven acute rejection episode at M12
To determine and compare according to randomized group | 12 months
  Graft and patient survival at M12
To determine and compare according to randomized group | 12 months
  Overall safety assessment

CONTACTS AND LOCATIONS:
Overall Officials: Yvon LEBRANCHU, Principal Investigator — University Hospital, Tours
Locations (16):
- France (16):
  - Hôpital Sud, Amiens
  - CHU de Angers, Angers
  - Hôpital Bois-Guillaume, Bois-Guillaume
  - Hôpital Cavale Blanche, Brest
  - CHU de Caen, Caen
  - Hôpital Gabriel Montpied, Clermont-Ferrand
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Hôpital Dupuytren, Limoges
  - Hôpital Archet II, Nice
  - HEGP, Paris
  - Hôpital Necker, Paris
  - Hôpital Maison Blanche, Reims
  - Hôpital Pontchaillou, Rennes
  - Hôpital Civil, Strasbourg
  - CHU de Toulouse, Toulouse
  - CHRU de Tours, Tours

REFERENCES:
- [Derived] Gatault P, Kamar N, Buchler M, Colosio C, Bertrand D, Durrbach A, Albano L, Rivalan J, Le Meur Y, Essig M, Bouvier N, Legendre C, Moulin B, Heng AE, Weestel PF, Sayegh J, Charpentier B, Rostaing L, Thervet E, Lebranchu Y. Reduction of Extended-Release Tacrolimus Dose in Low-Immunological-Risk Kidney Transplant Recipients Increases Risk of Rejection and Appearance of Donor-Specific Antibodies: A Randomized Study. Am J Transplant. 2017 May;17(5):1370-1379. doi: 10.1111/ajt.14109. Epub 2017 Jan 3. PMID 27862923